CLINICAL TRIAL: NCT05804006
Title: The Feasibility and Effects of Recumbent Cycling-based High-intensity Interval Training on Functional Performances, Cognitive Function, and Quality of Life in Early Subacute Stroke
Brief Title: High-Intensity Interval Training in the Early Subacute Stroke With a Semi-recumbent Bike
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hasselt University (Other)
Collaborators: Université de Parakou (Other)
Responsible Party: Principal Investigator, Dominique Hansen, Full Professor of Rehabilitation/Exercise Physiology in Cardiometabolic Diseases, Hasselt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0557CLERB-UP/P/SP/R/SA
Record Dates: First submitted 2023-02-15; First posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Stroke, Acute
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Conventional physiotherapy followed by High-Intensity Interval training on the semi-recumbent bike
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HIIT-REC (Experimental): High-intensity interval training program on a recumbent cycle SOLE R92 (HIIT-REC)
  Interventions: Other: Conventional physiotherapy followed by HIIT-REC program

INTERVENTIONS:
Other: Conventional physiotherapy followed by HIIT-REC program — The experimental protocol will be preceded by 30 minutes of conventional physiotherapy followed by 15 min the rest period; then the HIIT-REC procedure will start at 4-min at 30% of the peak workload interspersed with 1-min at 70% of the peak workload at 50 rpm for weeks 1-2 and increased by approximately 5 minutes every two weeks as tolerated to reach 30 minutes from week 5 (4 to 6 repetitions). The training intensity will progress similarly by 5% peak workload two weeks as tolerated to reach 4-min at 40% peak workload interspersed with 1-min 80% peak workload from week-5

SUMMARY:
Although High-intensity interval training (HIIT) exercise has emerged in recent years as a powerful time-efficient alternative to moderate-intensity continuous cardiovascular exercise training (MICT) to enhance neuroplasticity, motor, and cognitive functions, its feasibility remains to be determined early after stroke. Our study aims to investigate the feasibility of the HIIT program and its effects on functional abilities, cognitive function, and quality of life in early post-stroke.

DETAILED DESCRIPTION:
Study design, setting, and ethical considerations:

This study will be a prospective pre-post study that will be conducted at the university hospital of Parakou in Benin. The study protocol will be submitted to the ethics committee of Hasselt University in Belgium and the local biomedical ethics committee of the University of Parakou, Republic of Benin.

Interventions:

The experimental protocol will be preceded by 30 minutes of conventional physiotherapy, including neuromuscular interventions (balance training, postural awareness), musculoskeletal interventions (passive range of motion, stretching, strengthening), and lower-intensity overground walking. The conventional physiotherapy will be followed by 15 min of the rest period, then the experimental protocol consisting of a HIIT program on a recumbent cycle SOLE R92 (HIIT-REC) will be performed three times per week for six successive weeks.21 Training will be performed on non-consecutive days, thereby permitting recovery between sessions. The HIIT procedure will start at 4-min at 30% of the peak workload interspersed with 1-min at 70% of the peak workload at 50 rpm for weeks 1-2 and increased by approximately 5 minutes every two weeks as tolerated to reach 30 minutes from week 5 (4 to 6 repetitions). The training intensity will progress similarly by 5% peak workload two weeks as tolerated to reach 4-min at 40% peak workload interspersed with 1-min 80% peak workload from week-5.22 All sessions will be supervised and performed individually with verbal encouragement.

ELIGIBILITY:
Inclusion Criteria:

1. first episode from an ischemic or hemorrhagic stroke confirmed by CT scan;
2. muscular weakness of the leg on the hemiplegic side defined as NIHSS-Item 6 score between 1 and 3;
3. Ashworth score of 0 or 1, indicating no spasticity or slight spasticity over the affected lower limb, respectively
4. able to walk at least 5 meters independently with or without assistive devices and understand spoken instructions;
5. living in Parakou or the surrounding area and wishing to undergo the program at the hospital.

Exclusion Criteria:

Participants:

1. unable to perform a graded exercise test, i.e., unable to maintain the designated pedaling rate;
2. cardiovascular diseases (uncontrolled arrhythmias, decompensated heart failure or recent myocardial injury, arteriopathy);
3. primary orthopedic conditions (fractures, active rheumatoid arthritis);
4. other neurological diseases such as (Parkinson's disease and Alzheimer's disease).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility aspects | Up to 6 weeks
  The feasibility aspects, include recruitment rates (eligible population / consented population x 100), program adherence (attended sessions / total number of sessions x 100), and the safety (percentage of participants who will experience adverse events)
The change in the credibility of the treatment and the expectations of the participants | Week 1 and Week 6
  The treatment credibility and participant expectancy for improvement will be assessed with the Credibility and Expectancy Questionnaire (CEQ). The CEQ includes six items assessing a cognitively based credibility factor and an affectively based expectancy factor

SECONDARY OUTCOMES:
Berg Balance Scale | Week 1 and Week 6
  The Berg Balance Scale will be used to assess balance impairment. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function. The minimum score is 0 and the maximum score is 56. A score of 56 indicates functional balance and a score < 45 indicates a higher risk of falling.
5-Repetition Sit-To-Stand test | Week 1 and Week 6
  We will evaluate functional lower extremity strength with the 5-Repetition Sit-To-Stand test. The 5-Repetition Sit-To-Stand test measures the time taken to complete five repetitions of the sit-to-stand maneuver.
modified Rankin Scale | Week 1 and Week 6
  The modified Rankin Scale (mRS) will be used to evaluate the degree of disability in the daily activities. The mRS is an ordered scale coded from 0 (no symptoms at all) through 5 (severe disability)
6-min walk test | Week 1 and Week 6
  The 6-min walk test will be used to assess walking endurance. It assesses the distance a participant can walk as fast as possible for 6 min on a 30 m straight line with the option to stop for fatigue at any point.
10 m walk test | Week 1 and Week 6
  The 10mWT will be used to evaluate walking speed. It assesses the walking speed in meters per second over a short distance
Mini-Mental Stage Examination | Week 1 and Week 6
  The cognitive functions will be evaluated with the MMSE. It comprises thirty items providing information about orientation, attention, learning, calculation, delayed recall, and construction. The MMSE scores are interpreted as followed: > 25 (normal cognitive status), 18-23 (Mild cognitive impairment), and 0-17 (Severe cognitive impairment)
The 5-level EQ-5D version | Week 1 and Week 6
  We will use the EQ-5D-5L to assess the health-related quality of life (HRQoL). It comprises five health dimensions such as mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems

CONTACTS AND LOCATIONS:
Overall Officials: Oyene R Kossi, PhD, Study Director — University of Parakou; Thierry R Adoukonou, MD, PhD, Study Director — University of Parakou; Peter R Feys, PhD, Principal Investigator — Hasselt University
Locations (1):
- Faculty of Rehabilitation Sciences, Diepenbeek, Belgium

IPD SHARING:
Plan to Share IPD: No
Data will be available to researchers upon request to the first author (ERA)